CLINICAL TRIAL: NCT00581828
Title: Does Treatment of Hypovitaminosis D Increase Calcium Absorption?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0159; 05-1235-02
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Results first posted 2012-09-14 (Estimated); Last update posted 2023-07-24 (Actual); Status verified 2012-09

CONDITIONS: Osteoporosis; Osteopenia; Vitamin D Deficiency; Hypoparathyroidism; Hypercalciuria; Hypercalcemia
Keywords: Calcium Absorption; Intestinal Absorption of Calcium; Fractional Calcium Absorption; Stable Calcium Isotopes; Hypovitaminosis D; Vitamin D; Bone Mineral Density; Physical Function
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Vitamin D Deficiency; Hypoparathyroidism; Hypercalciuria; Hypercalcemia | interventions — Vitamin D; Ergocalciferols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Subjects received vitamin D (50,000 IU daily for 15 days) and maintenance dose vitamin D (50,000 IU twice monthly for 10 months).
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — 50,000 IU po qd for 15 days and 50,000 IU po twice month for 10 months (until final study visit at one year)
  Other Names: Vitamin D2; Ergocalciferol

SUMMARY:
The purpose is to perform a one-year study designed to assess whether treatment of hypovitaminosis D increases intestinal absorption of calcium, subsequent retention of calcium within bone, decreases bone turnover, and favorably impacts upon skeletal muscle mass, functional status, measures of physical function and quality of life. I hypothesize that treatment of hypovitaminosis D results in improved intestinal calcium absorption, greater retention of calcium within the bone reservoir and improved physical function, quality of life and muscle mass.

DETAILED DESCRIPTION:
Postmenopausal women with vitamin D insufficiency will participate in this one-year study. We will study the change in intestinal calcium absorption from baseline (vitamin D insufficiency) to follow up (vitamin D repletion and whether increased absorption results in subsequent increased retention of calcium within bone over the one-year interval as measured by bone densitometry. We will also study the effect of vitamin D repletion upon whole body muscle mass, quality of life and physical function.

A review of medical records and a screening visit will determine eligibility. Eligible and consenting subjects will present to the GCRC in the early morning and following baseline labs, will consume breakfast with a glass of orange juice enriched with a stable calcium isotope, and will receive 3 mg of another stable calcium isotope by intravenous injection. Over the next eight hours, blood will be taken a total of 9 more times and over the first 24 hours, all urine and stool will be collected for measurement of its calcium content.

Subsequently for the next five days, women will collect three urine specimens daily. Women will then receive vitamin D to treat vitamin D deficiency. Once vitamin D repletion is accomplished, all women will repeat their 24-hour visit and subsequent five-day urine collections. Women will maintain vitamin D repletion by taking a twice monthly tablet (50,000 IU) of vitamin D2. To confirm vitamin D repletion and safety over the full one year study, additional study visits will occur at 3, 6 and 12 months.

A bone density test at screening and twelve months will allow us to assess the effect of vitamin D repletion on whole body bone mass and skeletal mass. At each GCRC stay, 3, 6 and 12 months, women will complete questionnaires regarding quality of life and functional status and will perform the Timed Up and Go Test. Because we wish to maintain and confirm constant calcium intake throughout the one- year study, women will complete a calcium questionnaire at baseline, 3, 6 and 12 months.

With each subject's consent, we will collect one tube of blood and isolate its DNA. When sufficient knowledge is available regarding the pathophysiologic mechanisms whereby genetic polymorphisms impact calcium homeostasis, we will test for such DNA polymorphisms and relate genetic information with other data collected on calcium homeostasis.

ELIGIBILITY:
Inclusion Criteria:

* women at least five years past onset of menopause, defined as date of last menses (ages reported above are the range in ages of the participants recruited to the study)
* serum 25(OH)D 16-24 ng/ml by reverse phase HPLC
* calcium intake < or = 1,100 mg daily

Exclusion Criteria:

* Intake of >1,100 mg of calcium per day through the combination of diet and supplements
* Hypercalcemia (baseline serum calcium above the normal reference range)
* Nephrolithiasis, documented in the medical record or by patient report
* Inflammatory bowel disease, malabsorption, chronic diarrhea, or use of antibiotics within the past month
* Creatinine >2.0 mg/dL
* Hypercalciuria (baseline urine calcium: creatinine ratio >0.25)
* Current use of medications known to interfere with vitamin D and/or calcium metabolism, including oral steroids or anticonvulsants
* Ongoing or recent (past six months) use of bisphosphonates, estrogen compounds, calcitonin or teriparatide, as these compounds may independently affect retention of calcium within bone
* Diagnosis of, or evidence for, osteomalacia, manifest by serum 25(OH)D < 16 ng/ml or the presence of at least two of the following blood tests: low calcium, low phosphorus, or elevated alkaline phosphatase (23).
* Prior adult clinical fragility fracture or baseline T-score below -3.0 at the lumbar spine or femur

Ages: 50 Years to 66 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2005-01; Primary Completion 2008-07 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen E Hansen, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Background] Hansen KE, Jones AN, Lindstrom MJ, Davis LA, Engelke JA, Shafer MM. Vitamin D insufficiency: disease or no disease? J Bone Miner Res. 2008 Jul;23(7):1052-60. doi: 10.1359/jbmr.080230. PMID 18302509

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamin D: Subjects received vitamin D (50,000 IU daily for 15 days) and maintenance dose vitamin D (50,000 IU twice monthly for 10 months).
Period: Overall Study
Arm/Group | Vitamin D
Started | 19
Completed | 18
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vitamin D
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Intestinal Calcium Absorption From Baseline to One Month
Description: percent and true fractional calcium absorption
Time Frame: 1 month
Population: One subject's urine sample was mishandled, leaving 18 subjects with complete data for analysis.
Measure: Mean (Standard Deviation); unit: percent calcium absorption
Arm/Group | Vitamin D
Number analyzed (Participants) | 18
percent calcium absorption | 3 (1)

ADVERSE EVENTS:
Arm/Group | Vitamin D
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No